CLINICAL TRIAL: NCT02337764
Title: A Multicenter, Open-label, Long-term, Phase 3 Study to Evaluate the Safety and Efficacy of TVP-1012 at 1 mg in Levodopa Treated Parkinson's Disease Patients
Brief Title: A Long-term, Phase 3 Study of TVP-1012 (1 mg) in Levodopa Treated Parkinson's Disease Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TVP-1012/OCT-002; U1111-1165-1500 (Other: WHO); JapicCTI-152762 (Registry Identifier: JapicCTI)
Record Dates: First submitted 2015-01-09; First posted 2015-01-14 (Estimated); Results first posted 2019-04-19 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-02

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TVP-1012 1mg (Experimental): TVP-1012 1 mg once daily orally, either before or after breakfast, concomitantly with levodopa tablet for 52 weeks as treatment period after 2 weeks of run-in period.
  Interventions: Drug: TVP-1012 1mg

INTERVENTIONS:
Drug: TVP-1012 1mg — TVP-1012 1mg Tablets

SUMMARY:
The purpose of this study is to evaluate long-term safety of TVP-1012 (1 mg/day) with levodopa in Japanese participants with Parkinson's disease.

DETAILED DESCRIPTION:
This is a multicenter, open-label, long-term, phase 3 study to evaluate the safety and efficacy of long-term administration of TVP-1012 at 1 mg with levodopa in Japanese participants with Parkinson's disease.

The study period consisted of a 2-week run-in period and a subsequent 52-week treatment period. Participants fulfilling the inclusion criteria and did not meet any of the exclusion criteria at the start of the run-in period (Week -2) and also at the end of the run-in period (Week 0) were enrolled in the study, and received 1 mg of TVP-1012 once daily for 52 weeks, in an unblinded manner, from the day after Week 0.

ELIGIBILITY:
Inclusion Criteria:

* In the opinion of the investigator or sub-investigator, the participant is capable of understanding and complying with protocol requirements.
* The participant signs and dates a written, informed consent form and any required privacy authorization prior to the initiation of any study procedures.
* The participant has a diagnosis of Parkinson's disease according to the diagnostic criteria of the UK Parkinson's Disease Society Brain Bank.
* The participant has received a levodopa combination drug for >= 1 month at the start of the run-in period and has either of the following.

  * Wearing off phenomenon
  * Decreased response to levodopa combination drugs
* The participant has been receiving a levodopa combination drug a stable dose regimen since the start of the run-in period.
* The participant is an outpatient of either sex aged >= 30 and < 80 years at the time of consent.
* A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent to 1 month after the last dose of the investigational drug.

Exclusion Criteria:

* The participant has received any investigational medication within 90 days prior to the start of the run-in period.
* The participant has received TVP-1012 in the past.
* The participant is a study site employee, an immediate family member, or in a dependent relationship with a study site employee who is involved in the conduct of this study (e.g., spouse, parent, child, sibling) or may consent under duress.
* Participant has donated 400 mL or more of his or her blood volume within 90 days prior to the start of the run-in period.
* The participant has Modified Hoehn & Yahr stage 5 (or stage 5 at eather on-time or off-time for the participant with wearing off phenomenon) at the start of the run-in period.
* The participant has severe dyskinesia.
* The participant has unstable systemic disease.
* The participant has a Mini-Mental State Examinations (MMSE) score of <= 24 at the start of the run-in period..
* The participant has known or a history of schizophrenia, major or severe depression, or any other clinically significant psychiatric disease.
* The participant has a history of hypersensitivity or allergies to TVP-1012 (including any associated excipients) or selegiline.
* The participant has a history of clinically significant hypertension or other reactions associated with ingestion of tyramine-rich food (e.g., cheese, lever, herring, yeast, horsebean, banana, beer or wine).
* The participant has a history or concurrent of drug abuse or alcohol dependence.
* The participant has received neurosurgical intervention for Parkinson's disease (e.g., pallidotomy, thalamotomy, deep brain stimulation).
* The participant has received transcranial magnetic stimulation within 6 months prior to the start of the run-in period.
* The participant has received selegiline, pethidine, tramadol, reserpine or methyldopa within 90 days prior to the start of the run-in period.
* The participant has received single agent of levodopa, any psychoneurotic agent or antiemetic medication of dopamine agonist within 14 days prior to the start of the run-in period. However, the participant has been receiving quetiapine or domperidone with a stable dose regimen for >= 14 days prior to the start of the run-in period may be included in the study.
* The participant is required to take any of the prohibited concomitant medications or treatments.
* If female, the participant is pregnant or lactating or intending to become pregnant during, or within 1 month after the last administration of study medication in this study; or intending to donate ova during such time period.
* The participant has clinically significant neurologic, cardiovascular, pulmonary, hepatic (including mild cirrhosis), renal, metabolic, gastrointestinal, urological, endocrine, or hematological disease.
* The participant has clinically significant or unstable brain or cardiovascular disease, such as:

  * clinically significant arrhythmia or cardiac valvulopathy,
  * heart failure of NYHA Class II or higher,
  * concurrent or a history of ischemic cardiac disease within 6 months prior to the start of the run-in period,
  * concurrent or a history of clinically significant cerebrovascular disease within 6 months prior to the stat of the run-in period,
  * severe hypertension (systolic blood pressure of 180 mmHg or higher, or diastolic blood pressure of 110 mmHg or higher),
  * clinically significant orthostatic hypotension (including those with diastolic pressure decrease of 30 mmHg or more following postural change from supine/sitting position to standing position), or
  * a history of syncope due to hypotension within 2 years prior to the stat of the run-in period.
* The participant is required surgery or hospitalization for surgery during the study period.
* Participant has a history of cancer within 5 years prior to the start of the run-in period, except cervix carcinoma in situ which has completely cured.
* The participant has acquired immunodeficiency syndrome (AIDS) [including human immunodeficiency virus (HIV) carrier], or hepatitis [including viral hepatitis carrier such as hepatitis B surface (HBs) antigen or hepatitis C antibody (HCV) positive]. However, the participant who has a negative result for HCV antigen or HCV-RNA can be included in the study.
* The participant with laboratory data meeting any of the following at the start of the run-in period:

  * Creatinine >= 2 x upper limit of normal (ULN)
  * Total bilirubin >= 2 x ULN
  * ALT or AST >= 1.5 x ULN
  * ALP >= 3 x ULN
* The participant has received any of the prohibited concomitant medications or treatments during the run-in period
* The participant who, in the opinion of the investigator or sub-investigator, is unsuitable for any other reason.

Ages: 30 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2015-02-03 (Actual); Primary Completion 2016-09-29 (Actual); Study Completion 2016-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (24):
- Japan (24):
  - Nagoya, Aichi-ken
  - Matsuyama, Ehime
  - Fukuoka, Fukouka
  - Kōriyama, Fukushima
  - Sapporo, Hokkaido
  - Himeji, Hyōgo
  - Kobe, Hyōgo
  - Sanda, Hyōgo
  - Tsuchiura, Ibaragi
  - Ichinoseki, Iwate
  - Kawasaki, Kanagawa
  - Sagamihara, Kanagawa
  - Yokohama, Kanagawa
  - Tenri, Nara
  - Shimajiri-gun, Okinawa
  - Chuo-ku, Tokyo
  - Meguro-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Fukuoka
  - Kochi
  - Kyoto
  - Miyazaki
  - Osaka
  - Yamagata

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 25 investigative sites in Japan, from 03-Feb-2015 to 29-Sep-2016.
Pre-assignment Details: Participants with diagnosis of Parkinson's disease were enrolled in run- in period (Week -2 to 0). After that, the participants who fulfilled the inclusion criteria and did not meet any of the exclusion criteria at Week -2 and 0 were enrolled in the study and received TVP-1012 1 mg in an unblinded manner, from the day after Week 0.
Groups:
- TVP-1012 1 mg: For 2 weeks during the run-in period, followed by 52 weeks during the treatment period, TVP-1012 1 mg once daily orally, either before or after breakfast, concomitantly with levodopa tablet.
Period: Overall Study
Arm/Group | TVP-1012 1 mg
Started | 222
Completed | 162
Not Completed | 60
Not completed — Pretreatment Event/Adverse Event | 46
Not completed — Voluntary Withdrawal | 12
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set: All participants who received at least 1 dose of study drug.
Arm/Group | TVP-1012 1 mg
Number analyzed (Participants) | 222
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.0 (8.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 125
  Male | 97
Region of Enrollment [Number; unit: Participants]
  Japan | 222
Height [Mean (Standard Deviation); unit: centimeter (cm)] | 156.4 (9.67)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 55.86 (12.292)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/m^2 | 22.70 (3.821)
Smoking Classification [Number; unit: Participants]
  Current Smoker | 12
  Ex-Smoker | 80
  Never Smoked | 130
Timing of Study Drug Dose [Number; unit: Participants]
  Before Breakfast | 106
  After Breakfast | 116
Duration of Parkinson's Disease [Mean (Standard Deviation); unit: Years] | 7.09 (5.022)
Duration of Levodopa Use [Mean (Standard Deviation); unit: Years] | 4.61 (4.217)
Levodopa Total Daily Dose [Mean (Standard Deviation); unit: miligram (mg)] | 355.0 (147.11)
Levodopa Frequency per Day [Mean (Standard Deviation); unit: Times] | 3.3 (1.00)
Concomitant Use of COMT Inhibitor [Number; unit: Participants] — COMT; catechol-O-methyltransferase
  Participants
    Had COMT Inhibitor | 75
    Had no COMT Inhibitor | 147
Concomitant Use of Dopamine Agonist [Number; unit: Participants]
  Had Dopamine Agonist | 163
  Had no Dopamine Agonist | 59
Concomitant Use of Amantadine [Number; unit: Participants]
  Had Amantadine | 54
  Had no Amantadine | 168
Concomitant Use of Anticholinergics [Number; unit: Participants]
  Had Anticholinergics | 36
  Had no Anticholinergics | 186
Concomitant Use of Droxidopa [Number; unit: Participants]
  Had Droxidopa | 15
  Had no Droxidopa | 207
Concomitant Use of Istradefylline [Number; unit: Participants]
  Had Istradefylline | 26
  Had no Istradefylline | 196
Concomitant Use of Zonisamide [Number; unit: Participants]
  Had Zonisamide | 36
  Had no Zonisamide | 186
Wearing Off Phenomenon [Number; unit: Participants]
  Had Wearing Off Phenomenon | 116
  Had no Wearing Off Phenomenon | 106
Duration of Wearing Off Phenomenon [Mean (Standard Deviation); unit: Years] — Population: The number analyzed is the number of participants with data available for analysis.
  Years
    number analyzed (Participants) | 116
    (all) | 3.02 (2.747)
Modified Hoehn & Yahr Stage (ON State) [Mean (Standard Deviation); unit: Units on a scale] — Modified Hoehn & Yahr Stage represented severity for symptoms of Parkinson's disease progress. The Stage of Modified Hoehn & Yahr were assigned from Stage 0 (Asymptomatic) to Stage 5 (Wheelchair bound or bedridden unless aided (unable to walk even if aided)). Population: The number analyzed is the number of participants with data available for analysis.
  Units on a scale
    number analyzed (Participants) | 116
    (all) | 2.47 (0.688)
Modified Hoehn & Yahr Stage (OFF State) [Mean (Standard Deviation); unit: Units on a scale] — Population: The number analyzed is the number of participants with data available for analysis.
  Units on a scale
    number analyzed (Participants) | 116
    (all) | 3.19 (0.700)
Mean Daily OFF-time [Mean (Standard Deviation); unit: Hours] — Off-time refers to times when levodopa is not working well, causing worsening symptoms. Population: The number analyzed is the number of participants with data available for analysis.
  Hours
    number analyzed (Participants) | 111
    (all) | 4.99 (3.263)
Modified Hoehn & Yahr Stage [Mean (Standard Deviation); unit: Units on a scale] — Population: The number analyzed is the number of participants with data available for analysis.
  Units on a scale
    number analyzed (Participants) | 106
    (all) | 2.42 (0.708)
MDS-UPDRS Part II Total Score [Mean (Standard Deviation); unit: Scores on a scale] — Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) retained the 4-scale structure with a reorganization of the various subscales; (Part I) non-motor experiences of daily living (13 items), (Part II) motor experiences of daily living (13 items), (Part III) motor examination (33 scores based on 18 items), and (Part IV) motor complications (6 items). Each items had 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The scale range for Part II Total Score was 0-52, with higher scores reflecting greater severity.
  Scores on a scale | 11.9 (7.28)
MDS-UPDRS Part III Total Score [Mean (Standard Deviation); unit: Scores on a scale] — MDS-UPDRS retained the 4-scale structure with a reorganization of the various subscales; (Part I) non-motor experiences of daily living (13 items), (Part II) motor experiences of daily living (13 items), (Part III) motor examination (33 scores based on 18 items), and (Part IV) motor complications (6 items). Each items had 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The scale range for Part III Total Score was 0-132, with higher scores reflecting greater severity.
  Scores on a scale | 28.8 (13.14)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Experience at Least One Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs)
Time Frame: Up to Week 52
Population: Safety Analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | TVP-1012 1 mg
Number analyzed (Participants) | 222
Participants
  TEAEs | 185
  SAEs | 39

2. Secondary Outcome: Number of Participants With TEAE Related to Clinical Laboratory Tests
Time Frame: Up to Week 52
Population: Safety Analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | TVP-1012 1 mg
Number analyzed (Participants) | 222
Participants
  Blood creatine phosphokinase increased | 7
  Gamma-glutamyltransferase increased | 4
  Blood alkaline phosphatase increased | 3
  Blood lactate dehydrogenase increased | 1
  Blood uric acid increased | 1
  Liver function test value increased | 1
  Urine ketone body present | 1

3. Secondary Outcome: Number of Participants With Markedly Abnormal Vital Signs Values
Time Frame: Up to Week 52
Population: Safety Analysis set included all participants who received at least 1 dose of study drug. Here number of participants analyzed are participants evaluable for this outcome measure.
Measure: Number; unit: Participants
Arm/Group | TVP-1012 1 mg
Number analyzed (Participants) | 221
Participants
  Temperature (<35.6 °C) | 40
  Temperature(>37.7 °C) | 4
  Systolic Blood Pressure (<90 mmHg) | 33
  Systolic Blood Pressure (>180 mmHg) | 6
  Diastolic Blood Pressure(<50 mmHg) | 31
  Diastolic Blood Pressure (>100 mmHg) | 6
  Pulse (<45 bpm) | 1

4. Secondary Outcome: Number of Participants With TEAE Related to Electrocardiograms (ECG)
Time Frame: Up to Week 52
Population: Safety Analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | TVP-1012 1 mg
Number analyzed (Participants) | 222
Participants
  Atrial fibrillation | 3
  Supraventricular extrasystoles | 1

5. Secondary Outcome: Number of Participants With TEAE Related to Body Weight (Weight Decreased)
Time Frame: Up to Week 52
Population: Safety Analysis set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: Participants
Arm/Group | TVP-1012 1 mg
Number analyzed (Participants) | 222
Participants | 1

6. Secondary Outcome: Change From Baseline in Movement Disorder Society-Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II Total Score
Description: Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) retained the four-scale structure with a reorganization of the various subscales; (Part I) non-motor experiences of daily living (13 items), (Part II) motor experiences of daily living (13 items), (Part III) motor examination (33 scores based on 18 items), and (Part IV) motor complications (6 items). Each items had 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The scale range for Part II Total Score was 0-52, with higher scores reflecting greater severity.
Time Frame: Baseline and Week 52 (LOCF)
Population: Full Analysis Set included all participants who received at least 1 dose of the study drug. Here number of participants analyzed are participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TVP-1012 1 mg
Number analyzed (Participants) | 218
Units on a scale | 0.0 (5.08)

7. Secondary Outcome: Change From Baseline in MDS-UPDRS Part III Total Score
Description: Movement Disorder Society-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) retained the four-scale structure with a reorganization of the various subscales; (Part I) non-motor experiences of daily living (13 items), (Part II) motor experiences of daily living (13 items), (Part III) motor examination (33 scores based on 18 items), and (Part IV) motor complications (6 items). Each items had 0-4 ratings, where 0 = normal, 1 = slight, 2 = mild, 3 = moderate, and 4 = severe. The scale range for Part III Total Score was 0-132, with higher scores reflecting greater severity.
Time Frame: Baseline and Week 52 (LOCF)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | TVP-1012 1 mg
Number analyzed (Participants) | 215
Units on a scale | -7.6 (10.45)

8. Secondary Outcome: Change From Baseline to Week 52 (LOCF) in Mean Daily OFF-time
Description: Off-time refers to times when levodopa is not working well, causing worsening symptoms.
Time Frame: Baseline and Week 52 (LOCF)
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | TVP-1012 1 mg
Number analyzed (Participants) | 106
Hours | -0.89 (2.537)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | TVP-1012 1 mg
Serious Adverse Events (participants affected / at risk) | 39/222
Other Adverse Events (participants affected / at risk) | 81/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TVP-1012 1 mg (N=222)
Acute myocardial infarction (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Cataract (Eye disorders) | 1
Retinal detachment (Eye disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Large intestine polyp (Gastrointestinal disorders) | 1
Rectal prolapse (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Decreased activity (General disorders) | 1
Pyrexia (General disorders) | 1
Bacterial infection (Infections and infestations) | 1
Gastroenteritis norovirus (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 3
Femur fracture (Injury, poisoning and procedural complications) | 2
Spinal compression fracture (Injury, poisoning and procedural complications) | 2
Contusion (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fractured sacrum (Injury, poisoning and procedural complications) | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1
Rib fracture (Injury, poisoning and procedural complications) | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Parkinson's disease (Nervous system disorders) | 1
Parkinsonian gait (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Hallucination (Psychiatric disorders) | 1
Hallucination, visual (Psychiatric disorders) | 1
Psychiatric symptom (Psychiatric disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1
Aortic dissection (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | TVP-1012 1 mg (N=222)
Nasopharyngitis (Infections and infestations) | 31
Fall (Injury, poisoning and procedural complications) | 37
Contusion (Injury, poisoning and procedural complications) | 18
Dyskinesia (Nervous system disorders) | 24
Orthostatic hypotension (Vascular disorders) | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.